CLINICAL TRIAL: NCT06711211
Title: A Descriptive, Multicentre, Observational Epidemiological Study on Digestive Tumours
Brief Title: Spanish Registry of Digestive Tumours RETUD
Acronym: RETUD
Status: Recruiting | Type: Observational
Sponsor: Spanish Cooperative Group for the Treatment of Digestive Tumours (TTD) (Other)
Responsible Party: Sponsor
Other Study IDs: TTD-20-01 RETUD RETUD
Record Dates: First submitted 2024-11-25; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Digestive Cancers; Bile Duct Cancer; Hepatocellular Cancer (HCC); Colorectal Cancer (CRC); Pancreatic Cancer; Rectal Cancer
Keywords: digestive; cancer; tumours; cholangiocarcinoma; hepatocellular; colorectal; pancreas; rectal
MeSH Terms: conditions — Gastrointestinal Neoplasms; Bile Duct Neoplasms; Liver Neoplasms; Colorectal Neoplasms; Pancreatic Neoplasms; Rectal Neoplasms; Neoplasms; Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — * Frozen or formalin-fixed and paraffin-embedded tumour tissue samples, primary or metastatic, to be accompanied whenever possible by frozen or formalin-fixed and paraffin-embedded non-tumour tissue from the patient.
  * Liquid samples: Blood for obtaining serum and plasma.
  * By-products derived from these samples, such as circulating free DNA, circulating tumour cells, DNA, RNA, proteins, etc.
  Samples are obtained from patients undergoing surgery and/or from biopsies for diagnosis or treatment of the digestive tumours specified, always as part of the health care provided to them.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Biliary Tract Cancer (BTC): Patients diagnosed with cholangiocarcinoma or gallbladder carcinoma from 01-01-2017.
- Hepatocellular Carcinoma (HCC): Patients with hepatocellular carcinoma primary diagnosed from 01-01-2017 and treated with systemic therapy.
- MSI-High Colorectal Cancer (MSI-H CRC): Patients with MSI-High colorectal cancer (by PCR or IHQ) and primary pathological diagnosis from 01-01-2017.
- Pancreatic Cancer: Patients with exocrine pancreatic cancer diagnosed from 01-01-2019.
- Rectal Cancer: Patients diagnosed with rectal cancer from 01-01-2019.

SUMMARY:
The aim of this observational study is to assess the current state of digestive tumours in Spain. By doing so, it seeks to enhance the quality of care, optimize the diagnosis and treatment of digestive tumours, and identify opportunities for improvement that can benefit patients.

The study will investigate the epidemiological, biological, and clinical characteristics of digestive tumors diagnosed in patients aged 18 and older across healthcare centres in Spain. It also aims to generate knowledge and scientific evidence for events and situations that may impact on patients with digestive tumours (e.g. COVID-19 coronavirus pandemic).

Furthermore, subject to the patient's consent, biological samples may be collected for use in translational research projects and for the identification of molecular markers that may be useful in healthcare decision-making.

DETAILED DESCRIPTION:
Data will be collected ambispectively, recording those patients who were diagnosed with digestive tumours before the start of the study (from 2017) and also those who are diagnosed after the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥18 years old diagnosed with oesophageal cancer, gastric cancer, pancreatic cancer, hepatocarcinoma, gallbladder and bile duct cancer, cancer of the small intestine, appendix and gastrointestinal stroma, colorectal cancer, anal canal cancer or digestive hereditary cancer.
* Written informed consent available.

Exclusion Criteria:

* Patient for whom, for whatever reason, it is not possible to know or obtain the information necessary to complete the data collection base.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with digestive tumours in healthcare centres of Spain.
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2020-12-23 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Situation of digestive tumours in Spain | For each cohort, an annual data cut-off (12 months) is planned. Epidemiology, therapy and efficacy parameters are analyzed from date of diagnosis to outcome or cut-off date, for registry population (at least baseline visit completed)
  Understanding the situation of digestive tumours in Spain, their epidemiology (risk factors, age, sex), biology and clinical manifestations in order to improve the quality of care, optimise diagnosis and treatment, and identify areas for improvement that can benefit patients.

SECONDARY OUTCOMES:
Knowledge about situations that can impact digestive tumours | An annual data cut-off (12 months) per cohort is planned. Upon specific situations (i.e COVID-19), specific cohorts are open to capture related data
  Generate knowledge and scientific evidence on events and situations that may impact on digestive tumours (e.g. COVID-19 coronavirus pandemic).
Biological substudies for translational reseach of tumor diagestive diseases | Frequency of translational projects is defined for each indivial substudy, with data captured from firts´subject diagnosis to last subject´s outcome at time of database
  Subjects may consent in translational projects (i.e. biomarkers determination, NGS or DNA analysis, etc), with banked biological samples
Determination of molecular markers | Frequency of translational projects is defined for each indivial substudy, with data captured from firts´subject diagnosis to last subject´s outcome at time of database
  Determination of molecular markers that may be useful healthcare decision-making in patients diagnosed with digestive tumours.

CONTACTS AND LOCATIONS:
Locations (1):
- Grupo de Tratamiento de los Tumores Digestivos (TTD), Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication or a presentation to a scientific congress or meeting
Supporting Information: Study Protocol, ICF, CSR
Time Frame: At cohort interim analysis, regularly, average of one update per year
Access Criteria: Abstracts, posters, oral presentation to congresses, scientific publication related to RETUD patient cohort analysis, will be shared by statisticians, authors, contributors and referees involved in publication peer-review.